CLINICAL TRIAL: NCT06976489
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Crossover Study to Evaluate the Food Effect on the Safety and the Pharmacokinetics of PA-111 in Healthy Adult Volunteers
Brief Title: The Food Effect on PK Characteristics and Safety Profiles of PA-111
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PA-111FE
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Mixed Dyslipidemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: Fasted, Period 2: Fed
  Interventions: Drug: PA-111
- Sequence B (Experimental): Period 1: Fed, Period 2: Fasted
  Interventions: Drug: PA-111

INTERVENTIONS:
Drug: PA-111 — PA-111 1Tab., Per Oral

SUMMARY:
Primary endpoint of this study is to evaluate the pharmacokinetic characteristics of PA-111 in healthy subjects.

DETAILED DESCRIPTION:
The purpose of this study is to compare and evaluate the effect of food on the safety and pharmacokinetic profiles of PA-111 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight equal to or greater than 50kg (Female 45kg) and Body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2 at the time of screening visit
* The Age equal to or greater than 19 in healthy volunteers at the time of screening visit

Exclusion Criteria:

* Participation in another clinical study with an investigational drug within the 6 months from scheduled first administration
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration of drug in plasma (Cmax) | pre-dose (0hour) to 72hours
  Cmax of PA-111
Area under the plasma concentration-time curve during dosing interval (AUCt) | pre-dose (0hour) to 72hours
  AUCt of PA-111

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No